CLINICAL TRIAL: NCT02440984
Title: Anorectal Dysfunction in Patients Suffering From Spina Bifida : From Clinic to Neuro-epithelial Function
Brief Title: Anorectal Dysfunction in Patients Suffering From Spina Bifida : From Clinic to Neuro-epithelial Function (ANOSPIN)
Acronym: ANOSPIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015-A00082-47; 35RC15_8926 (Other: CHU Rennes)
Record Dates: First submitted 2015-04-28; First posted 2015-05-12 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Spina Bifida
Keywords: enteric nervous system; anorectal disorder; barostat anorectal; physiology; spina bifida
MeSH Terms: conditions — Spinal Dysraphism; Rectal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Enteric nervous system dysfunction (Other): colonic biopsies and usual care
  Interventions: Procedure: Colonic biopsies during endoscopy

INTERVENTIONS:
Procedure: Colonic biopsies during endoscopy — eligible patients will have physical examination, colonic biopsies during endoscopy and anal manometry with barostat. these investigations are part of the usual healthcare. Colonic biopsies will be used to study intestinal permeability, colonic inflammation and enteric nervous system.

SUMMARY:
The purpose of this study is to assess and explain (at least apart) anorectal disorders of patients with Spina Bifida by an automatic neuropathy responsive of enteric nervous system and epithelial barrier dysfunctions. The investigators' aim hypothetics is that autonomic neuropathy of patients with Spina Bifida induce enteric nervous sytem and epithelial barrier dysfunctions which explain anorectal disorders of these patients. Thexpect to show a decreased of 5% of enteric neurons per ganglia.

DETAILED DESCRIPTION:
Spina Bifida is rare disease related to a failure of the closure of neural tube during the embryonic period. This malformation results in a variety of clinical disorders (neurologic, urologic, orthopedic, anorectal), depending on the level of the spinal cord lesion. Anorectal functional disorders remain underestimated and unknown from a pathophysiological point of view with subsequent uncodified therapeutic strategy.

Patients with Spina Bifida always present autonomic neuropathy that contributes partially to the anorectal disorders. These disorders may be related to a closed relationship between autonomic and enteric nervous system. Both nervous systems play a key role in anorectal disorders during others neurological disaeses have a common and simultaneous development from neural crest and induce colonic epithelial changes related to the closed connection between epithelial barrier and enteric nervous system. All of this remains hypothetic because no data regarding the impairment of enteric nervous system and epithelial barrier are available and no study are ongoing on this topic.

ELIGIBILITY:
Inclusion Criteria:

* patient aged between 18 and 65 years old
* patient who consulted to the national Spina Bifida Center for multidisciplinary assessment or for a proctology/urologic clinic
* need of colonic biopsies during endoscopy
* free, written and informed consent

Exclusion Criteria:

* pregnancy or breastfeeding
* protected adults (judicial protection, guardianship and truesteeship) and persons deprived of liberty
* patient unable to giving their consent
* anticoagulants therapy or coagulation disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-06-15 (Actual); Primary Completion 2019-06-15 (Estimated); Study Completion 2019-12-15 (Estimated)

PRIMARY OUTCOMES:
number of enteric neurons per ganglia | data collected at the day of endoscopy
  all data will be collected in the Spina Bifida database for further analyses. Colonic biopsies will be used to study intestinal permeability, colonic inflammation and enteric nervous system

SECONDARY OUTCOMES:
anorectal symptoms | data collected at the day of endoscopy
Rectal compliance | data collected at the day of endoscopy
  Rectal compliance is defined by a volume variation during ascending pressure (phasic distension). It will be performed with a bag connected to electronic barostat.
Likert scale | data collected at the day of endoscopy
  Sensation intensity will be measured at each pressure step, by using 6-point Likert scale ranging from 0 (no sensation) to 6 (intolerable pain)
macroscopic and microscopic colonic inflammation | data collected at the day of endoscopy
intestinal permeability marker | data collected at the day of endoscopy
  Intestinal permeability will be measured using Ussing chamber.
number of glia cells per ganglia | data collected at the day of endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Charlène Brochard, Md, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, France

REFERENCES:
- [Derived] Brochard C, Bouguen G, Olivier R, Durand T, Henno S, Peyronnet B, Pagenault M, Lefevre C, Boudry G, Croyal M, Fautrel A, Esvan M, Ropert A, Dariel A, Siproudhis L, Neunlist M. Altered epithelial barrier functions in the colon of patients with spina bifida. Sci Rep. 2022 May 3;12(1):7196. doi: 10.1038/s41598-022-11289-3. PMID 35505001